CLINICAL TRIAL: NCT06157541
Title: Phase I/II Clinical Trial of Allogeneic Cytomegalovirus-specific T Cells in Combination With Pembrolizumab for Recurrent and Newly Diagnosed Glioblastoma Multiforme
Brief Title: T Cells and Pembrolizumab for Recurrent and Newly Diagnosed Glioblastoma
Acronym: TCaP
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Queensland Institute of Medical Research (Other)
Collaborators: CUREator (Unknown); Merck Sharp & Dohme LLC (Industry); The Newro Foundation (Unknown); Royal Brisbane and Women's Hospital (Other Government); Princess Alexandra Hospital, Brisbane, Australia (Other); Austin Hospital, Melbourne Australia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: P3894 / MSD-MK3475-E78
Record Dates: First submitted 2023-11-26; First posted 2023-12-06 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Glioblastoma Multiforme; Astrocytoma, Grade IV
Keywords: immunotherapy; T cells; pembrolizumab; glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Phase I of the trial is a 3+3 dose escalation study involving 9-18 participants. Phase II will recruit two cohorts of 20 participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Part 1 (Experimental): Patients with recurrent disease. Interventions:
  * allogeneic CMV-specific T cells (cell suspension for infusion), dose cohorts: 2 × 10^7 cells, 4 × 10^7 cells, 8 × 10^7 cells; 4 infusions; administered weekly
  * pembrolizumab 400 mg (solution for injection); 18 infusions; administered every 6 weeks
  Interventions: Biological: Allogeneic cytomegalovirus-specific T cells; Drug: Pembrolizumab
- Part 2 Group A (Experimental): Patients with recurrent disease. Interventions:
  * allogeneic CMV-specific T cells (cell suspension for infusion), maximum-tolerated dose identified in phase I; 4 infusions; administered weekly
  * pembrolizumab 400 mg (solution for injection); 18 infusions; administered every 6 weeks
  Interventions: Biological: Allogeneic cytomegalovirus-specific T cells; Drug: Pembrolizumab
- Part 2 Group B (Experimental): Patients with newly diagnosed disease. Interventions:
  * allogeneic CMV-specific T cells (cell suspension for infusion), maximum-tolerated dose identified in phase I; 4 infusions; administered weekly
  * pembrolizumab 400 mg (solution for injection); 18 infusions; administered every 6 weeks
  Interventions: Biological: Allogeneic cytomegalovirus-specific T cells; Drug: Pembrolizumab

INTERVENTIONS:
Biological: Allogeneic cytomegalovirus-specific T cells — Allogeneic cytomegalovirus (CMV)-specific T cells generated from the blood of healthy CMV-seropositive donors
  Other Names: CYT-101
Drug: Pembrolizumab — A humanised immunoglobulin G4 (IgG4) monoclonal antibody (mAb) specific for the programmed cell death 1 (PD-1) receptor
  Other Names: Keytruda

SUMMARY:
The goal of this clinical trial is to test a combined therapy approach (allogeneic cytomegalovirus [CMV]-specific T cells and pembrolizumab) in patients with brain cancer. The type of brain cancer being studied is glioblastoma multiforme/astrocytoma grade 4.

The purpose of part 1 of this study is to determine the maximum-tolerated dose and/or recommended dose(s) for future exploration of allogeneic CMV-specific T cells as monotherapy or in combination with pembrolizumab in patients with recurrent GBM/astrocytoma grade 4. Part 2 of the study aims to investigate the anti-tumour activity of allogeneic CMV-specific T cells as monotherapy or in combination with pembrolizumab, assessed by magnetic resonance imaging and survival, in patients with recurrent or newly diagnosed GBM/grade 4 astrocytoma.

DETAILED DESCRIPTION:
This is a multi-centre, non-randomised, open-label, dose escalation and expansion trial of allogeneic cytomegalovirus (CMV)-specific T cells as monotherapy and in combination with pembrolizumab in participants with recurrent and newly diagnosed glioblastoma multiforme (GBM)/astrocytoma grade 4. The trial will be conducted in two parts.

Part 1 is a single-arm, sequential 3+3 dose-escalation of allogeneic CMV-specific T cells as a monotherapy and in combination with a fixed dose of pembrolizumab to determine the recommended dose(s) for future exploration. Up to 18 participants will be recruited for part 1. Part 2 will involve two arms and will examine the clinical impact of the CMV-specific T cells as monotherapy and in combination with pembrolizumab. Forty participants will be recruited for part 2 - 20 with newly diagnosed GBM/astrocytoma grade 4 and 20 with recurrent GBM/astrocytoma grade 4.

Part 2 will only be initiated if the data and safety monitoring board (DSMB) determines that the proposed dose level(s) for future exploration are safe and well tolerated. Additional groups may be explored depending on emergent safety, pharmacodynamics and/or clinical efficacy data.

Following screening and enrolment, each participant will receive four weekly infusions (Q1W) of allogeneic CMV-specific T cells, followed by up to 18 infusions of pembrolizumab. Pembrolizumab infusions will commence seven days (±3 days) after the final T-cell infusion, and be administered every 6 weeks (Q6W). The total duration of participation for each participant is approximately 26 months.

Efficacy of the combination therapy will be evaluated according to the modified Response Assessment in Neuro-Oncology (RANO) and immunotherapy (i)RANO criteria, through radiographic imaging. For group A and group B the appropriate measures for progression-free survival (PFS), overall survival (OS), disease control rate and duration of response will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age on the day of signing informed consent, with histologically confirmed diagnosis of GBM or astrocytoma Grade 4^.

   a. For participants with recurrent GBM or astrocytoma grade 4, histological confirmation of primary diagnosis is available i. First occurrence of disease progression with radiological confirmation ≥12 weeks from completion of radiation therapy.

   ii. Where surgical resection of recurrent disease occurred, histological confirmation of GBM or astrocytoma Grade 4 is required.

   b. For participants with newly diagnosed GBM or astrocytoma Grade 4, histological confirmation of diagnosis is required i. Participant, in consultation with their treating clinicians, is willing to delay the commencement of standard of care adjuvant temozolomide until the completion of CMV-specific T cell therapy infusions.

   ^Note: Histological confirmation using the 2016 or 2021 World Health Organization (WHO) Classification of Tumours of the central nervous system (CNS) is acceptable and classification edition will be noted.
2. Male participants: Must agree to use contraception during the treatment period and for at least 180 days after the last dose of study treatment and refrain from donating sperm during this period.
3. Female participants: Must not be pregnant or undergoing in vitro fertilisation or breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) OR
   2. A WOCBP who agrees to follow contraceptive guidance during the treatment period and for at 120 days after the last dose of study treatment.
4. Provision of written informed consent for the trial. Approved interpreters will be used for patients who do not have sufficient understanding of English for informed consent to be obtained without an interpreter.
5. Participants who have AEs due to previous anti-cancer therapies must have recovered to ≤Grade 1 or baseline. Participants with endocrine-related AEs who are adequately treated with hormone replacement or participants who have ≤Grade 2 neuropathy are eligible. Participants with >Grade 1 adverse events (AEs) due to previous anti-cancer therapies may be allowed to enrol on a case-by-case basis in discussion with the study Sponsor, if it is determined that it will not put the participant at a higher risk of study-related AEs or interfere with the integrity of the study outcome.
6. For participants with disease progression, this should be the first evidence of measureable disease based on modified RANO criteria. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
7. CMV-positive serology
8. Provision of consent for the use of archival formalin-fixed, paraffin embedded or fresh tumour tissue obtained at the time of surgical resection or excisional biopsy.
9. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
10. Have a life expectancy of at least 6 months.
11. Have adequate organ function. Specimens must be collected within 10 days prior to the start of study intervention.
12. Have availability of an human leukocyte antigen (HLA)-matched batch of allogeneic CMV-specific T cells.
13. Provision of consent to access to Medicare Benefits Schedule (MBS) and Pharmaceutical Benefits Scheme (PBS) patient/provider health information collected by Services Australia (phase II participants only).
14. Criteria for known hepatitis B and C positive participants:

Hepatitis B and C screening tests are not required unless:

* Known history of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* As mandated by local health authority

14.1 Hepatitis B-positive participants:

* Participants who are HBsAg positive are eligible if they have received HBV anti-viral therapy for at least 4 weeks and have undetectable HBV viral load prior to enrolment.
* Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention

14.2 Participants with history of HCV infection are eligible if HCV viral load is undetectable at screening.

• Participants must have completed curative anti-viral therapy at least 4 weeks prior to enrolment.

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to the first dose of study intervention (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor.
3. Has received prior systemic anti-cancer therapy or investigational agents within 4 weeks prior to study intervention, with the exception of temozolomide, which is permitted during the trial.
4. Recurrent disease cohorts only: Has not yet recovered from all radiation-related toxicities not requiring corticosteroids other than dexamethasone, or has had radiation pneumonitis.

   Note: A 1-week washout is permitted for palliative radiation of non-CNS disease (≤2 weeks of radiotherapy). Participants receiving dexamethasone must be clinically stable and receiving a stable or weaning dose of ≤2 mg/day 1-2 weeks prior to the commencement of pembrolizumab.
5. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study intervention. Administration of killed vaccines is allowed.
6. Has received in an investigational agent, or has used an investigational device within 4 weeks prior to the first dose of study intervention.
7. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
8. Known additional malignancy that is progressing or has required active treatment within the past 5 years.

   Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, prostate cancer treated with radical prostatectomy, or carcinoma in situ, excluding carcinoma in situ of the bladder, who have undergone potentially curative therapy are not excluded. Participants with additional malignancy within the past 5 years may be allowed to enrol on a case-by-case basis, in discussion with the study Sponsor, if the malignancy is deemed of very low recurrence potential and the participant has completed curative intent therapy.
9. Has a previous known GBM/astrocytoma grade 4 recurrence previously treated with surgery, radiotherapy and/or chemotherapy, and evidence of further progression or recurrence.
10. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid).
12. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
13. Has an active infection requiring systemic therapy.
14. Has a known history of human immunodeficiency virus (HIV) infection. Note: No HIV testing is required unless mandated by a local health authority.
15. Concurrent active hepatitis B (defined as HBsAg positive and/or detectable HBV DNA) and hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection.

    Note: Hepatitis B and C screening tests are not required unless:
    * Known history of HBV and HCV infection
    * As mandated by local health authority
16. Has not adequately recovered from major surgery or has ongoing surgical complications.
17. Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
18. Has known psychiatric or substance-abuse disorders that would interfere with cooperation with the requirements of the trial.
19. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
20. Has had an allogeneic tissue/solid organ transplant or stem cell transplant.
21. Has a baseline corrected QT interval (QTc) of >450 ms, assessed by ECG. If the participant's screening ECG records a QTc of >450 ms, the ECG is to be done in triplicate and the average of the QTc is to be recorded. If the QTc remains >450 ms, the participant will be excluded from enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities | Within 49 days of receiving the first dose of study drug
  Part 1 - Primary Endpoint 1
Incidence of adverse events and clinically significant changes in laboratory parameters, vital signs, and electrocardiograms (ECGs) | Within 49 days of the first dose of study drug
  Part 1 - Primary Endpoint 2
Percentage of participants with confirmed complete response (CR) or partial response (PR) | Within 25 months of the first dose of study drug
  Part 2 - Primary Endpoint 1
Percentage of participants with confirmed complete response (CR), partial response (PR), or stable disease (SD) | Within 25 months of the first dose of study drug
  Part 2 - Primary Endpoint 2
Duration of response | Within 25 months of the first dose of study drug
  Part 2 - Primary Endpoint 3
Overall survival (percentage of participants alive) | 6 months
  Part 2 - Primary Endpoint 4
Progression-free survival (percentage of participants with no evidence of further disease progression) | 6 months
  Part 2 - Primary Endpoint 5

SECONDARY OUTCOMES:
Percentage of participants with confirmed CR or PR | Within 25 months of the first dose of study drug
  Part 1 - Secondary Endpoint 1
Percentage of participants with confirmed CR, PR, or SD | Within 25 months of the first dose of study drug
  Part 1 - Secondary Endpoint 2
Duration of response | Within 25 months of the first dose of study drug
  Part 1 - Secondary Endpoint 3
Overall survival (percentage of participants alive) | 6 months
  Part 1 - Secondary Endpoint 4
Progression-free survival (percentage of participants with no evidence of further disease progression) | 6 months
  Part 1 - Secondary Endpoint 5
Incidence of adverse events and clinically significant changes in laboratory parameters, vital signs, and ECGs | Within 25 months of the first dose of study drug
  Part 2 - Secondary Endpoint 1

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Khanna, PhD, Principal Investigator — QIMR Berghofer Medical Research Institute
Locations (4):
- Australia (4):
  - Newro Foundation, Bowen Hills, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Austin Hospital, Heidelberg, Victoria

IPD SHARING:
Plan to Share IPD: No